CLINICAL TRIAL: NCT00405340
Title: Rituximab in the Treatment of Idiopathic Membranous Nephropathy
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Fernando Fervenza, M.D., Ph.D., Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-004833
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Membranous Nephropathy
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Rituximab

ARMS (1):
- Drug (Experimental): Rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Patients will received rituximab 4 weekly doses of rituximab 375 mg/m2 at baseline. Patients will be retreated at 6 months.

SUMMARY:
Membranous glomerulopathy (MN) is still the most common glomerular disease associated with nephrotic proteinuria (NS). Up to 40% of patients reach end stage renal failure (ESRD), making MN the 2nd or 3rd most common cause of ESRD caused by a primary glomerulopathy. Current treatment options include corticosteroids, alkylating agents, and cyclosporin, but their use is controversial and the associated adverse effects and high cost temper their usage. Experimental data in MN suggests that B cell activation results in immunoglobulin deposition along the glomerular basement membrane causing injury to the membrane and subsequent proteinuria. Drugs that non-selectively inhibit B cells and, these pathogenic antibodies, are closely associated with improved outcomes. Based on the rationale that selective depletion of B cells in humans would prevent the production of ?nephrotoxic? immunoglobulins and subsequent renal injury we recently treated 15 patients with MN with rituximab 1g i.v. twice (day 1 and day 15). Baseline proteinuria of 13.0±5.5g/24h decreased to 9.1±7g, 9.7±8g and 6.5±6 g/24h at 3, 6, and 9 months, respectively (mean ± SD). Analysis of the pharmacokinetic data obtained from this study, however, suggests that in heavily nephrotic patients, rituximab dosed in this fashion results in patients being under-treated. The present study propose to test the hypothesis that rituximab, given in accordance to the standard lymphoma protocol (375mg/m2 x 4), will result in a more effective and profound depletion of B cells, a more complete suppression of pathogenic antibodies, and a higher remission rate of the NS while maintaining a favorable safety profile.

DETAILED DESCRIPTION:
a. Study Overview: Once a patient with idiopathic MN and proteinuria >5g/24h is identified and meets other entry criteria, he/she will receive a minimum of 4 months of non-immunosuppressive therapy aimed at maximizing Ang II blockade (run-in phase). The target blood pressure (<130 mmHg systolic BP >75% of the readings; but not <100 mmHg systolic) is chosen based on recent recommendations by the JNC VII.(38) 1) The first step will be the administration of an ARB. This is chosen because ARBs are as effective as ACEIs in blocking the AT1 mediated adverse effects of Ang II, while being better tolerated, with minimal cough or angioedema, and less hyperkalemia. Because this part of the study aims to maximize Ang II blockade, ARB dose will continue to be increased every 2 weeks until the maximum tolerated/FDA approved dose is achieved or until intolerable side effects occur (e.g. development of postural hypotension, light headed, hyperkalemia, etc). 2) Once ARB dose has been maximize and there are no observable side-effects, and/or blood pressure is not at target, a long acting ACEi will be added. ACEi dose will be increased every 2 weeks aiming to achieve maximum tolerated or maximum approved dosage. For patients whose blood pressure control is not at target additional medication will be added in the following order: 3) a loop diuretic, 4) a cardioselective β-blocker, 5) a non-dihydropyridine calcium channel blocker (CCB), and 6) clonidine. The selection of these drugs adheres to the recommendation of the JNC VII.(38) The choice of a non-dihydropyridine CCB was made because of concerns that dihydropyridine-type CCB may obscure the anti-proteinuric effects of the above therapy. In order to further ensure that any potential adverse effect is minimized we have limited CCB to be used as a fifth agent, and to be used only when the combination of ARB/ACEi, diuretic, and β-blocker have failed to reduce BP to target level. Concomitant Treatment: 1. At the start of the run-in/conservative phase of the study, and as part of the standard of care for patients with NS and severe hyperlipidemia, patients will be started on atorvastatin 10 mg a day (or its equivalent) and if tolerated (no evidence of persistent elevation of liver transaminase >3x upper limit of normal, muscle pain, high CK, or rhabdomyolysis) the dose can be increased according to the recently published KDOQI-dyslipidemia guidelines.(39) The dose should not be increased above the maximum of 40 mg/day. The rationale for not using a higher statin dose is because of the risk of developing proteinuria with the use of statins at high doses. Patients will remain at the highest tolerated dose for the entire duration of the study. Serum lipids will be measured at baseline and every 3 months thereafter. 2. High sodium intake (e.g. >200 mm NaCl/d or 4.6 g sodium/d) can significantly impair the beneficial effects of Ang II blockade.(40) Therefore patients will be instructed to go on a low salt diet (2-3g/day). 3. Patients will receive dietary counseling at enrollment regarding a dietary protein target intake of 0.8 g/kg ideal body weight/day of high quality protein and will be encouraged to maintain the same diet throughout the duration of the study.

Rituximab: If at the end of this period the patient still meets entry criteria he/she will be treated with rituximab, 375 mg/m2 i.v. on days 1, 8, 15 and 22, with subsequent follow-up of at least one year. Patients will be retreated at month 6th once B-cells return to circulation and will be independent of the clinical status of the patient. B-cell return is defined as CD19+B cell count > 15/microliter or >5% of baseline count. There will be a +/- 3 day window for each study visit, to account for weekends, holidays, and scheduling conflicts.

Figure 3. Schematic time-line for the study. Primary endpoint.

1. Change in proteinuria from baseline to 12 months. This approach was selected taking in consideration that B cell recovery following administration of rituximab usually begins at 6 months after the last infusion, but it is not complete until 9-12 months later, (complete recovery is defined as normalization of CD19+ B cell counts; normal CD19+ count is 71-567 cells/μl).

Secondary endpoints.

1. Complete and partial remission rates at 6, 9, and 12 months (see definitions in Table 3)
2. Pharmacokinetics/bioavailability
3. Rate of decline in urinary protein
4. Frequency of relapse after CR
5. Toxicity

ELIGIBILITY:
* Idiopathic MN with diagnostic biopsy performed within the past 24 months.
* Age > 18 years
* If female, must be post-menopausal, surgically sterile or practicing a medically approved method of contraception
* Patients need to be treated with an ACEI and/or ARB, for at least 4 months prior to rituximab treatment and have adequately controlled blood pressure (BP <130/75 mm Hg in >75% of the readings).
* Proteinuria as measured by urinary proteinuria / urinary creatinine > 5.0 on a spot sample aliquot from a 24-hour urine collection.
* Estimated GFR ≥ 30 ml/min/1.73m2 while taking ACEI/ARB therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2010-07 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Primary endpoint. | 12 months

SECONDARY OUTCOMES:
Complete and partial remission rates at 6, 9, and 12 months | 6, 9, and 12 months
Pharmacokinetics/bioavailability | 12 months
Rate of decline in urinary protein | 12 months
Frequency of relapse after CR | 12 months
Toxicity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fernando C. Fervenza, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States